CLINICAL TRIAL: NCT05707390
Title: A Phase 1, Multicenter, Open-label, Single-dose Study to Assess the Pharmacokinetics of Mezigdomide in Healthy Participants and Those With Mild, Moderate, and Severe Hepatic Impairment
Brief Title: A Study of Mezigdomide in Healthy Participants and Participants With Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA057-1010
Record Dates: First submitted 2023-01-23; First posted 2023-01-31 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Hepatic Impairment
Keywords: Mezigdomide; BMS-986348; CC-92480

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Mild hepatic impairment (Experimental)
  Interventions: Drug: Mezigdomide
- Moderate hepatic impairment (Experimental)
  Interventions: Drug: Mezigdomide
- Severe hepatic impairment (Experimental)
  Interventions: Drug: Mezigdomide
- Healthy participants (Experimental)
  Interventions: Drug: Mezigdomide

INTERVENTIONS:
Drug: Mezigdomide — Specified dose on specified days
  Other Names: BMS-986348; CC-92480

SUMMARY:
The aim of this study is to measure the concentration levels of mezigdomide in the blood of participants with mild, moderate, and severe hepatic impairment, and in matched healthy control participants with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

Hepatic Impaired Participants:

* Participants have mild, moderate, or severe hepatic impairment or cirrhosis due to chronic hepatic disease and/or prior alcohol use.
* Participants have mild (Group A), moderate (Group B), or severe (Group C) hepatic impairment as defined by Child-Pugh Score.

Matched Healthy Participants:

* Participant must be free of any clinically significant disease that would interfere with the study evaluations.
* Participant must have liver-related laboratory test results within the respective reference ranges or with clinically insignificant excursions therefrom as agreed by the investigator.

Exclusion Criteria:

All Participants:

* History of chronic pruritus or dermatologic syndromes that may be confounded with reactions to mezigdomide.
* Contraindication or intolerance to first-generation antihistamine medications.

Hepatic Impaired Participants:

-Clinical laboratory test results:

* Platelet count lower than 30,000/microliter (μL) at screening or Day -1.
* Absolute neutrophil counts lower than 1,500/μL at screening or Day -1.

Matched Healthy Participants:

-History of or suspected benign ethnic neutropenia.

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) | Up to 6 days
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUC[0-T]) | Up to 6 days
Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUC[INF]) | Up to 6 days

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 6 days
Number of participants with serious adverse events (SAEs) | Up to 6 days
Number of participants with physical examination abnormalities | Up to 6 days
Number of participants with vital sign abnormalities | Up to 6 days
Number of participants with electrocardiogram (ECG) abnormalities | Up to 6 days
Number of participants with clinical laboratory abnormalities | Up to 6 days
Metabolic ratio of AUC(0-T) | Up to 6 days
Metabolic ratio of AUC(0-INF) | Up to 6 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (3):
  - PANAX, Miami Lakes, Florida
  - Orlando Clinical Research Center OCRC, Orlando, Florida
  - The Texas Liver Institute, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/content/studyconnect/us/en/clinical-trials/NCT05707390.html